CLINICAL TRIAL: NCT01560338
Title: Impact of Hypothermia on Midazolam and Morphine Pharmacokinetics
Brief Title: Hypothermia's Impact on Pharmacology
Acronym: HIP
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 12-009214; RO1HL11274501A1 (Other: NIHLBI)
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Cardiac Arrest; Hypothermia
Keywords: Pharmacokinetics; Midazolam; Morphine; Cardiac Arrest; Hypothermia
MeSH Terms: conditions — Heart Arrest; Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric after Cardiac Arrest: Pediatric patients greater than 3 kg. and less than 18 years suffering cardiac arrest who have been given or currently receiving morphine and/or midazolam and receiving hypothermia.

SUMMARY:
The purpose of the study will help us understand the complex interaction between hypothermia (cooling) and pharmacogenetics (how specific genes effect how drugs are handled), and their impact on how routinely given sedation drug are broken down and used by the body when given to children after cardiac arrest (when heart stops pumping blood) and are critically ill.

DETAILED DESCRIPTION:
Background:

Therapeutic hypothermia is used in the pediatric intensive care unit, and is being studied in the setting of pediatric cardiac arrest. Following cardiac arrest, multiple organ dysfunction syndrome, especially renal and hepatic dysfunction, is common and affects the metabolism and excretion of drugs. In addition, very little is known about the impact of hypothermia on a child's ability to metabolize medications. Dose adjustments may be required in the setting of hypothermia to avoid under-dosing and over-dosing of medications. Improper dosing and drug accumulation of sedatives and opiates can worsen existing neurologic, circulatory and respiratory failure. The measurement of the actual drug and metabolite concentrations in the body (pharmacokinetics) provides information on how a child metabolizes medications. In addition, variability in these concentrations after the administration of equal doses to different children may result from genetically driven differences in drug metabolizing systems (pharmacogenetics). Finally, these genetic differences may respond differently to hypothermia. Our overarching hypothesis is that morphine and midazolam disposition will be affected by temperature management even when accounting for potentially confounding quantifiable factors of organ dysfunction and genetic differences.

Objectives:

The objectives of this study, Hypothermia's Impact on Pharmacology 2, are

1. To estimate the impact of hypothermia on the variability in morphine and midazolam pharmacokinetics in children after cardiac arrest and
2. To estimate the impact of genetic factors on the variability in morphine and midazolam pharmacokinetics, specifically in the setting of hypothermia.

Sophisticated modeling and simulation techniques will be utilized to examine the highly dynamic changes in physiology associated with critical illness, drug disposition, pharmacogenetics and temperature modulation. The models created using this approach will be implemented to optimize the prospective treatment of these critically ill children.

Study Design:

Prospective pharmacokinetic study

ELIGIBILITY:
Inclusion Criteria:

* Be greater than or equal to three (3) kg
* Receiving or have received morphine and/or midazolam as part of clinical care
* Receiving hypothermia after any cardiac arrest
* Provide Informed Consent

Exclusion Criteria:

* Receiving renal replacement therapy [example Continuous Veno-Venous Hemofiltration (CVVH), Continuous Veno-Venous Hemodialysis (CVVHD), and Continuous Veno-Venous Hemodiafiltration (CVVHDF)]
* Receiving plasmapheresis

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population is the pediatric population equal to or greater than 3 kg and less than 18 years of age AND have had or currently receiving morphine and/or midazolam AND receive hypothermia after cardiac arrest administered as part of clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01-28 (Actual)

PRIMARY OUTCOMES:
Physiologic manifestations of cardiac arrest and Multiple Organ Dysfunction Syndrome (MODS) in relation to morphine and midazolam | 2.5 years
  The objective of this aim is to identify the physiologic manifestations of cardiac arrest and MODS that underlie the variability in morphine and midazolam pharmacokinetics.

SECONDARY OUTCOMES:
Impact of genetic factors | 2.5 years
  The objective of this aim is to estimate the impact of genetic factors that underlie the variability in morphine and midazolam pharmacokinetics (PK), specifically in the setting of pediatric cardiac arrest. In this aim we will investigate the effect of genotype on pharmacokinetic parameters for morphine and midazolam.

OTHER OUTCOMES:
Manifestations of hypothermia | 2.5 years
  The objective of this aim is to identify the manifestations of hypothermia that underlie the variability in morphine and midazolam pharmacokinetics in children after cardiac arrest. In this aim we will investigate the effect of body temperature on PK parameters for morphine and midazolam.

CONTACTS AND LOCATIONS:
Overall Officials: Athena F Zuppa, MD MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Louisville, Louisville, Kentucky
  - Univeristy of Michigan, Ann Arbor, Michigan
  - Nationwide Children's Medical Center, Columbus, Ohio
  - Pennsylvania State University Hersey Medical Center, Hershey, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided